CLINICAL TRIAL: NCT06517849
Title: The Stanford Gambling Addiction Therapy Study (SGATS) in Colorado
Brief Title: Beliefs About Mental Health Treatment - Gambling Addiction Study in Colorado
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Kindbridge Research Institute (Unknown)
Responsible Party: Principal Investigator, Sarah Bogl, Graduate Student, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 75109
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Gambling Disorder; Gambling Problem; Mental Health Issue
Keywords: Beliefs; Bias; Incentive
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Intervention Model Description: Participants in the control group will take two (paid) surveys and have access to free cognitive behavioral therapy (CBT). Participants in the treatment group will be offered an additional payment (in the form of gift cards) to undergo a certain number of CBT sessions with Kindbridge Behavioral Health.
Who Masked: Care Provider
Masking Description: Participants will know whether they are offered the incentive or not. Care providers (i.e., counselors at Kindbridge Behavioral Health) will not know (and participants can access care regardless of whether they are in the treatment group or not).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Incentive (No Intervention): The "No Incentive" arm will participate in two surveys-including questions about beliefs about therapy and willingness to pay for therapy, gambling behavior, and well-being-at the baseline and at the end (four months after the first survey). The arm will have access to free cognitive behavioral therapy through Kindbridge Behavioral Health, but will not receive a monetary incentive to undergo therapy.
- Fixed Incentive (Experimental): The "Fixed Incentive" arm will participate in two surveys-including questions about beliefs about therapy and willingness to pay for therapy, gambling behavior, and well-being-at the baseline and at the end (four months after the first survey). The arm will have access to free cognitive behavioral therapy through Kindbridge Behavioral Health and will be offered a modest monetary incentive to undergo therapy. The incentive will be in form of an electronic gift card. The amount of money offered as an incentive will not depend on the participants' survey replies.
  Interventions: Behavioral: Monetary Incentive for Take-Up of Cognitive Behavioral Therapy
- Payment According to Multiple Price List Choices (Experimental): The "Multiple Price List" arm will participate in two surveys-including questions about beliefs about therapy and willingness to pay for therapy, gambling behavior, and well-being-at the baseline and at the end. The arm will have access to free cognitive behavioral therapy through Kindbridge Behavioral Health and might be offered a modest monetary incentive to undergo therapy. More specifically, for all arms, the surveys will include a multiple price list to gauge willingness to pay for CBT. For this "multiple price list" arm, one of the rows from the multiple price list will be (randomly) picked and implemented. Depending on what the participant answered in the randomly picked row, they will either receive an unconditional payment or a payment conditional on undergoing CBT. In either case, the payment will be in form of an electronic gift card.
  Interventions: Behavioral: Monetary Incentive for Take-Up of Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Monetary Incentive for Take-Up of Cognitive Behavioral Therapy — Both treatment arms will be offered a monetary incentive (in form of a retail gift card) for undergoing a certain number of CBT sessions.
  Arms: Fixed Incentive; Payment According to Multiple Price List Choices

SUMMARY:
Many people with mental health conditions do not seek treatment, and it is unclear what exactly prevents people from taking up treatment. The goal of this interventional study is to learn about how people think about cognitive behavioral therapy (CBT) for gambling disorders. The main questions it aims to answer are:

* Do people have incorrect beliefs about the net benefits of CBT? If yes, which beliefs are those, and how much do people underestimate or overestimate the benefits?
* Is a small monetary incentive (that participants receive conditional on trying out CBT) helpful in increasing take-up of CBT?

Apart from these questions, the researchers will also study how well CBT works to treat gambling disorders.

Participants will be asked to complete two surveys over four months and might be offered a modest monetary incentive for doing (free) CBT if they are in the treatment group. Researchers will compare that treatment group to a control group. Participants in the control group will have access to free CBT and do the same two surveys as those in the treatment group, but will not receive the monetary incentive.

ELIGIBILITY:
Inclusion Criteria:

* must reside in Colorado
* must be English-speaking

Exclusion Criteria:

* does not reside in Colorado
* is not English-speaking

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Willingness to Pay for CBT | Baseline and 4 months
  Change in participants' willingness to pay (in USD; elicited through multiple price lists) for CBT from baseline to follow-up survey.
Change in Beliefs about CBT | Baseline and 4 months
  Change in participants' beliefs about therapy (such as effectiveness, unpleasantness, stigma, etc.) will between baseline and follow-up survey (4 months after baseline).
Attendance of CBT sessions | 4 months
  Dates and number of CBT sessions participants attend (as long as they are with Kindbridge Behavioral Health) between baseline survey and follow-up survey (afer 4 months).
Change in Gambling Consumption | Baseline and 4 months
  Amount wagered (in USD) in online and offline gambling by participants over the last month. Difference between stated amount at baseline and stated amount in follow-up survey.
Change in Subjective Well-Being | Baseline and 4 months
  Change in measure of participants' wellbeing from baseline to follow-up (at four months), computed using Likert scale style questions about feeling happy/depressed/satisfied/anxious/etc. Answers are on a seven-point scale from "strongly disagree" through "neutral" to "strongly agree." Points for each question are coded such that more positive answers get more points (so from most negative to most positive, the points -1, -2/3, -1/3, 0, 1/3, 2/3, 1 are awarded) and subjective well-being is the sum of all points.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bogl, Principal Investigator — Stanford University; Matt Brown, Principal Investigator — Stanford University; Mariana Guido, Principal Investigator — Stanford University; Nick Grasley, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No